CLINICAL TRIAL: NCT04723498
Title: Problematic Use of the Internet in Child and Adolescent Psychiatry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Susanne Walitza (Other)
Responsible Party: Sponsor-Investigator, Susanne Walitza, Head of the Department of Child and Adolescent Psychiatry, Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KJPP 2020-00117
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Other): male and female patients, handled on an ambulatory basis in Psychiatric University Clinics, Department of Child and Adolescent Psychiatrythe ages from 8 - 18 years during the study
  Interventions: Diagnostic Test: screening questionnaire

INTERVENTIONS:
Diagnostic Test: screening questionnaire — Fill in screening questionnaire

SUMMARY:
Pathological internet use is a blanket term for problematic behavior types (e.g. uncontrolled gaming, cyber pornography, cyber mobbing and excessive use of social media): all perpetrated through the internet. There is little documentation or research on interdependencies/interplay between problematic internet and/or media use and child-adolescent disturbances. Very few clinical examples of syndromes like attention deficiency/hyperactivity (ADHS), anxiety disorder or affective disturbances associated with pathological media/internet use, or gaming, are found in literature.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients ages from 8 - 18 years
* All study participants or their legal representative have given written permission for their experiences to be documented in the study.

Exclusion Criteria:

* Inability to understand explanations and the questionnaire, whether linguistic or cognitative

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Symptoms severity of problematic internet and media use | 3 months
  The clinician screening questionnaire (PUI) contains 9 items designed to assess severity of problematic internet and media use of obsessive and compulsive in children and adolescents.The test uses a 4-point scale to rate severity of problematic internet and media use. Higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Walitza, Prof. Dr. med. Dipl.-Psych., Principal Investigator — Sponsor GmbH
Locations (1):
- Psychiatric University Clinics, Department of Child and Adolescent Psychiatry, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided